CLINICAL TRIAL: NCT03589014
Title: Treat_CCM Clinical Trial A Multicenter Randomized Clinical Trial on Propranolol in Familial Cerebral Cavernous Malformation
Brief Title: Treat_CCM: Propranolol in Familial Cerebral Cavernous Malformation
Acronym: Treat_CCM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: IFOM ETS - The AIRC Institute of Molecular Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRFMN-7358; 2017-003595-30 (EudraCT Number)
Record Dates: First submitted 2018-05-17; First posted 2018-07-17 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Cerebral Cavernous Malformation
Keywords: Cerebral Cavernous Malformation; Propranolol; Magnetic Resonance Imaging
MeSH Terms: conditions — Hemangioma, Cavernous, Central Nervous System | interventions — Propranolol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Treat_CCM is a Prospective Randomized Open Trial with Blinded Evaluation of outcomes (PROBE).
  Clinical events CCM-related (i.e. intra-cerebral hemorrhage and focal neurological deficits excluding seizures) will be blindly adjudicated by an independent Event Committee.All MRI exams will be read in a Central Laboratory by experienced neuroradiologists, unaware of patient identification and study treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard Treatments recommended for CCM
- ￼Propranolol (Experimental): Initial oral dose 40 mg bid, uptitrated to 80mg bid doses as low as 10 mg bid and up to 160 mg bid, 20 to 320mg daily, are acceptable according to tolerability.
  Interventions: Drug: Propranolol

INTERVENTIONS:
Drug: Propranolol — Patients randomized to the experimental arm will receive propranolol on top of standard recommended treatment for CCM. Initial oral dose of 40 mg bid will be uptitrated to 80 mg bid in the absence of excessive bradycardia or hypotension. Doses as low as 10 mg bid and up to 160 mg bid, 20 to 320mg daily, are acceptable according to tolerability.
  Other Names: Inderal
  Arms: ￼Propranolol

SUMMARY:
Cerebral Cavernous Malformation (CCM) is a cerebrovascular disease which can be either congenital in origin or sporadic and is characterized by the presence of isolated or multiple CCM lesions, causing recurrent headache, seizures, focal neurological deficits and hemorrhages. Inasmuch, to date, the only curative treatment available is limited to surgical lesion eradication or stereotactic radiosurgery. It is therefore necessary to find an effective medical treatment that may limit disease progression and decrease the burden of adverse clinical events. The non-selective betablocker propranolol has been found to be effective in the treatment of infantile cutaneous hemangioma, and anecdotal reports have been published on its efficacy in CCM. The safety profile of propranolol has been documented in millions of patients of all ages.

The primary objective of this exploratory trial is to test whether a chronic treatment with propranolol will reduce the burden of cerebrovascular lesions, of clinical events and symptoms in patients with familial CCM.

DETAILED DESCRIPTION:
The project will consist of a multicenter, open-label, randomized study (PROBE design) in patients with CCM to be randomized in a 2:1 ratio (propranolol:control) and will allow comparison of 2 groups: one receiving propranolol (recommended initial dose is 40 mg bid, to be uptitrated to 80 mg bid, however, doses as low as 10 mg bid and up to 160 mg bid are acceptable according to tolerability) on the top of recommended standard care, the other receiving recommended standard care. This investigator-driven study will be open-label with a PROBE design will be applied so that each MRI exam will be centrally read and all adverse clinical events will be centrally adjudicated. It should be pointed out that by no means surgery, whenever indicated, will be delayed and/or avoided because of study treatment allocation.

The purpose of this exploratory trial is to test whether a chronic treatment with propranolol will reduce the burden of cerebrovascular lesions, of clinical events and symptoms in patients with familial CCM. Inherited CCM is a rare disease with a prevalence of less than 5/10.000. Thus, since the number of patients to be included in this exploratory trial will be insufficient to prove or disprove a statistically significant beneficial effect of propranolol on clinical events, the extension to more centers and patients is formally included in the present protocol. Special care will be paid to the biologic consistency of the different endpoints, even if none of them will yield statistically significant differences. The assessment of the tolerability of propranolol in normotensive otherwise healthy patients is another clinically relevant endpoint.

If the overall evaluation of the safety (no difference in AEs and SAEs between propranolol and control arms), and of the efficacy profile (assessed as consistency between incidence of adverse clinical events and magnetic resonance brain imaging results between propranolol and control arms) at the conclusion of the present study, will be reassuring for propranolol, a protocol for a definitive Phase 2 trial will be submitted for approval to Regulatory Authorities. This second trial may be designed as single-arm as far as adequate data on incidence of endpoint events will be available from Treat_CCM.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Familial cerebral cavernous malformations (FCCM);
2. history of clinical symptoms or events: intracerebral hemorrhage, stroke, permanent or transient focal deficits, seizures, disability or any other neurological symptom supposedly related to CCM;
3. age of at least 18 years.
4. Written informed consent to participate in the study prior to any study procedures.

Exclusion Criteria:

1. Implanted pacemaker or any other condition preventing the magnetic resonance imaging (MRI);
2. bradycardia (<50 bpm) or 2nd or 3rd degree AV block, hypotension (symptomatic);
3. unstable diabetes;
4. severe asthma;
5. renal and/or liver failure;
6. current use of verapamil and diltiazem for risk of excessive bradycardia;
7. previous brain surgery (within 6 months);
8. known hypersensitivity to study drug (propranolol or any of the ingredients)
9. pregnant or lactating women or women of childbearing potential who are not protected from pregnancy by an accepted method of contraception
10. participation to another clinical trial;
11. inability to cooperate with the trial procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Adverse clinical events CCM-related. | up to 24 months
  New occurrence of clinical events CCM-related, that is intra-cerebral hemorrhage (ICH) and focal neurological deficits (FND) excluding seizures.

SECONDARY OUTCOMES:
De novo CCM lesions depiction on MRI. | up to 24 months
  De novo CCM lesions depiction will be obtained on MRI QSM and Susceptibility Weighted Images (SWI) that is very sensitive to hemoglobin and iron deposition.
Adverse clinical outcomes, other than ICH and FND. | up to 24 months
  Global disability and health related quality of life as assessed by Beck Depression Inventory -BDI- questionnaire. BDI is made of 21 questions scored on a scale from 0 to 3, 0 representing the best condition. Final score will be the sum of all scores and will range from 0 to 63, were 0 is the best condition. SF-36 is made of 36 questions scored on a scale from 0 to 100 representing the highest level of functioning possible. Questions are aggregated in 8 dimensions of health (eg pain, phsical functioning etc.).
Location and MRI signal characteristics of CCM lesions at MRI. | up to 24 months
  Location and MRI signal characteristics of CCM lesions will be assessed by 3 T brain MRI. The encephalic regions evaluated will be: cerebellum, brainstem, right/left hemisphere, right/left basal ganglia. Lesions with previous surgical treatment will be excluded from imaging analysis
Diameter of CCM lesions at MRI. | up to 24 months
  Diameter will be assessed in millimeters.
Length of CCM lesions at MRI | up to 24 months
  Length will be assessed in millimeters.
Micro-hemorrhages at MRI. | up to 24 months
  Micro-hemorrhages will be assessed by magnetic susceptibility of the brain tissue, a biophysical property proportional to local iron content (quantitative susceptibility mapping, QSM). Unit of Measure of QSM is parts per million (ppm). Changes from baseline will be calculated.
Dynamic contrast enhanced permeability (DCEP) at MRI. | up to 24 months
  Cerebral vascular permeability will be assessed after injection of gadolinium at MRI by dynamic contrast enhanced permeability (DCEP) method. Changes from baseline will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabetta Dejana, Professor, Study Chair — IFOM ETS - The AIRC Institute of Molecular Oncology; Roberto Latini, Study Director — Istituto Di Ricerche Farmacologiche Mario Negri
Locations (6):
- Italy (6):
  - IRCCS Casa Sollievo della Sofferenza, San Giovanni Rotondo, FG
  - IRCCS Centro Neurolesi "Bonino Pulejo", Messina, ME
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Mi
  - Fond. IRCCS Ist. Naz. Neurologico Carlo Besta, Milan, MI
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, MI
  - Fondazione Policlinico Universitario "A. Gemelli", Roma, RM

IPD SHARING:
Plan to Share IPD: Yes
Locking of the trial data base, completion of main analyses, and submission for publication of the main study result are expected to take at least 14 months after last patient-last-visit date.
  Only clinical data relative to patients' characteristics and follow-up will be shared for each individual patient. Biohumoral and imaging data will be shared only after approval by the Steering Committee of the trial of a specific request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: By Dec 31st 2021 IPD will be made available.
Access Criteria: Free access for clinical data. Biohumoral and imaging data will be shared only after approval by the Steering Committee of the trial of a specific request.
URL: https://www.marionegri.it/dipartimenti/medicina-cardiovascolare

REFERENCES:
- [Background] Lampugnani MG, Malinverno M, Dejana E, Rudini N. Endothelial cell disease: emerging knowledge from cerebral cavernous malformations. Curr Opin Hematol. 2017 May;24(3):256-264. doi: 10.1097/MOH.0000000000000338. PMID 28212190
- [Background] Bravi L, Malinverno M, Pisati F, Rudini N, Cuttano R, Pallini R, Martini M, Larocca LM, Locatelli M, Levi V, Bertani GA, Dejana E, Lampugnani MG. Endothelial Cells Lining Sporadic Cerebral Cavernous Malformation Cavernomas Undergo Endothelial-to-Mesenchymal Transition. Stroke. 2016 Mar;47(3):886-90. doi: 10.1161/STROKEAHA.115.011867. Epub 2016 Feb 2. PMID 26839352
- [Background] Cuttano R, Rudini N, Bravi L, Corada M, Giampietro C, Papa E, Morini MF, Maddaluno L, Baeyens N, Adams RH, Jain MK, Owens GK, Schwartz M, Lampugnani MG, Dejana E. KLF4 is a key determinant in the development and progression of cerebral cavernous malformations. EMBO Mol Med. 2016 Jan 1;8(1):6-24. doi: 10.15252/emmm.201505433. PMID 26612856
- [Background] Marchi S, Corricelli M, Trapani E, Bravi L, Pittaro A, Delle Monache S, Ferroni L, Patergnani S, Missiroli S, Goitre L, Trabalzini L, Rimessi A, Giorgi C, Zavan B, Cassoni P, Dejana E, Retta SF, Pinton P. Defective autophagy is a key feature of cerebral cavernous malformations. EMBO Mol Med. 2015 Nov;7(11):1403-17. doi: 10.15252/emmm.201505316. PMID 26417067
- [Background] Maddaluno L, Rudini N, Cuttano R, Bravi L, Giampietro C, Corada M, Ferrarini L, Orsenigo F, Papa E, Boulday G, Tournier-Lasserve E, Chapon F, Richichi C, Retta SF, Lampugnani MG, Dejana E. EndMT contributes to the onset and progression of cerebral cavernous malformations. Nature. 2013 Jun 27;498(7455):492-6. doi: 10.1038/nature12207. Epub 2013 Jun 9. PMID 23748444
- [Background] Boulday G, Rudini N, Maddaluno L, Blecon A, Arnould M, Gaudric A, Chapon F, Adams RH, Dejana E, Tournier-Lasserve E. Developmental timing of CCM2 loss influences cerebral cavernous malformations in mice. J Exp Med. 2011 Aug 29;208(9):1835-47. doi: 10.1084/jem.20110571. Epub 2011 Aug 22. PMID 21859843
- [Background] Bravi L, Rudini N, Cuttano R, Giampietro C, Maddaluno L, Ferrarini L, Adams RH, Corada M, Boulday G, Tournier-Lasserve E, Dejana E, Lampugnani MG. Sulindac metabolites decrease cerebrovascular malformations in CCM3-knockout mice. Proc Natl Acad Sci U S A. 2015 Jul 7;112(27):8421-6. doi: 10.1073/pnas.1501352112. Epub 2015 Jun 24. PMID 26109568
- [Background] Gore AV, Lampugnani MG, Dye L, Dejana E, Weinstein BM. Combinatorial interaction between CCM pathway genes precipitates hemorrhagic stroke. Dis Model Mech. 2008 Nov-Dec;1(4-5):275-81. doi: 10.1242/dmm.000513. Epub 2008 Oct 28. PMID 19093037
- [Derived] Meessen JMTA, Abete-Fornara G, Zarino B, Castori M, Tassi L, Carriero MR, D'Alessandris QG, Al-Shahi Salman R, Blanda A, Nicolis EB, Novelli D, Caruana M, Vasami A, Lanfranconi S, Latini R. Patient-reported outcome measures in patients with familial cerebral cavernous malformations: results from the Treat_CCM trial. Front Neurol. 2024 Feb 14;15:1338941. doi: 10.3389/fneur.2024.1338941. eCollection 2024. PMID 38419711
- [Derived] Lanfranconi S, Scola E, Meessen JMTA, Pallini R, Bertani GA, Al-Shahi Salman R, Dejana E, Latini R; Treat_CCM Investigators. Safety and efficacy of propranolol for treatment of familial cerebral cavernous malformations (Treat_CCM): a randomised, open-label, blinded-endpoint, phase 2 pilot trial. Lancet Neurol. 2023 Jan;22(1):35-44. doi: 10.1016/S1474-4422(22)00409-4. Epub 2022 Nov 17. PMID 36403580
- [Derived] Lanfranconi S, Scola E, Bertani GA, Zarino B, Pallini R, d'Alessandris G, Mazzon E, Marino S, Carriero MR, Scelzo E, Farago G, Castori M, Fusco C, Petracca A, d'Agruma L, Tassi L, d'Orio P, Lampugnani MG, Nicolis EB, Vasami A, Novelli D, Torri V, Meessen JMTA, Al-Shahi Salman R, Dejana E, Latini R; Treat-CCM Investigators. Propranolol for familial cerebral cavernous malformation (Treat_CCM): study protocol for a randomized controlled pilot trial. Trials. 2020 May 12;21(1):401. doi: 10.1186/s13063-020-4202-x. PMID 32398113